CLINICAL TRIAL: NCT01131611
Title: Cognitive-Behavioral Based Physical Therapy: Improving Surgical Spine Outcomes
Brief Title: Cognitive-Behavioral Physical Therapy
Acronym: CBPT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Kristin Archer, Assistant Professor, Vanderbilt University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 100508
Record Dates: First submitted 2010-05-24; First posted 2010-05-27 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Spinal Stenosis
Keywords: Spinal Stenosis; Rehabilitation; Physical Therapy (specialty); Cognitive Behavior Therapy; Behavioral Research
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBPT intervention (Experimental): Standard PT treatment + CBPT
  Interventions: Behavioral: CBPT
- Control-Attention (Placebo Comparator): Standard PT treatment + weekly phone calls
  Interventions: Other: Control-Attention

INTERVENTIONS:
Behavioral: CBPT — Cognitive-Behavioral Based Physical Therapy
  Arms: CBPT intervention
Other: Control-Attention — Standard of Care + weekly phone calls
  Arms: Control-Attention

SUMMARY:
The overall objective of this application is to conduct a two-group randomized controlled trial (RCT) to gather preliminary evidence on the efficacy of a brief cognitive-behavioral based PT (CBPT) intervention in patients at-risk for poor outcomes following lumbar spine surgery for degenerative conditions. Our central hypothesis is that incorporating cognitive and behavioral strategies into postoperative standard of care PT will improve surgical outcomes, through reductions in fear of movement and pain catastrophizing. We have established the feasibility of training therapists in the CBPT intervention, recruiting and retaining patients, and the procedures for data collection and study management. The long-term goal is to broaden the availability of well-accepted and effective CBT strategies by expanding the implementation from traditional providers, psychologists, to a group of providers, physical therapists, who routinely interact with musculoskeletal pain populations.

DETAILED DESCRIPTION:
Despite surgical advances, up to 40% of patients continue to have chronic pain and functional disability after lumbar spine surgery. Our own data demonstrate that high fear of movement is a risk factor for increased pain and disability in this patient population. Cognitive-behavioral therapy (CBT) and physical therapy (PT) interventions targeting fear of movement have proven effective for decreasing persistent pain and functional disability in patients with chronic low back pain. However, the efficacy of a combined CBT and PT approach has not been well demonstrated in a surgical spine population. Therefore, we propose to conduct a two-group randomized controlled trial (RCT) to gather preliminary evidence on the efficacy of a brief cognitive-behavioral based PT (CBPT) intervention in patients at-risk for poor outcomes following lumbar spine surgery for degenerative conditions. We hypothesize that incorporating cognitive and behavioral strategies into postoperative standard of care PT will improve self-reported pain and disability and observed physical function, through reductions in fear of movement and pain catastrophizing (i.e., tendency to magnify pain sensations). This pilot study plans to recruit 80 patients with high postoperative fear of movement or pain catastrophizing. These eligible at-risk patients will be randomized to one of the two groups: (1) standard PT treatment + CBPT or (2) standard PT treatment + weekly phone calls to control for attention. The CBPT program consists of 1 in person and 5 telephone sessions and is based on well-accepted and effective CBT strategies. These strategies focus on relaxation, problem-solving training, cognitive restructuring, and behavioral self management. Primary outcomes include self-reported pain and disability as measured by the Brief Pain Inventory and the Oswestry Disability Index. Secondary outcomes consist of observed physical function as measured by performance-based tests of gait speed, balance, repeated chair stands, and mobility (Short Physical Performance Battery, Timed Up and Go). Outcome data will be collected at baseline (6 weeks after surgery), after treatment (3 months after surgery), and at 6 months following surgery. The proposed two-group RCT will provide estimates of effect sizes and sample sizes associated with the CBPT intervention and data on feasible recruitment and retention goals and the mechanisms through which the CBPT intervention affects long-term outcomes. This informative pilot data will guide a multicenter, three-group clinical trial to further validate the CBPT intervention. Our long-term objective is to broaden the availability of effective CBT strategies by expanding the implementation from traditional providers, psychologists, to a group of providers, physical therapists, who routinely interact with a large population of patients with musculoskeletal pain.

ELIGIBILITY:
English speaking adults of both sexes and all races scheduled for lumbar spine surgery for a degenerative condition (spinal stenosis, spondylosis with or without myelopathy, and spondylolisthesis) will be considered for study participation.

Inclusion criteria will include the following:

1. Radiographic evidence of lumbar spinal stenosis secondary to degenerative changes;
2. Surgical treatment using laminectomy with or without arthrodesis (i.e., fusion);
3. Presence of back and/or lower extremity pain > 6 months;
4. No history of neurological movement disorder;
5. No presence of psychotic disease; and
6. TSK score > 39

Exclusion criteria will include the following:

1. Patients having microsurgical techniques as the primary procedure, such as an isolated laminotomy or microdiscectomy (individuals having these minimally invasive surgical techniques tend to have a less severe case of lumbar degeneration and a shorter recovery time than individuals having arthrodesis or laminectomy without arthrodesis);
2. Patients having surgery for spinal deformity as the primary indication (patients with spinal deformity as the primary spinal disorder tend to have a different recovery trajectory compared to the inclusion population); and
3. Patients having surgery secondary to pseudarthrosis, trauma, infection, or tumor.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | 6 months post-discharge from therapy
  The ODI measures disability

SECONDARY OUTCOMES:
Brief Pain Inventory (BPI) | 6 months post-discharge from therapy
  The BPI measures pain intensity and pain interference

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Archer, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Orthopaedic Institute, Nashville, Tennessee, United States